CLINICAL TRIAL: NCT02403011
Title: A Randomized Controlled Study in the Efficiency of Soft Tissue Mobilization in Babies With Congenital Muscular Torticollis and Deformational Plagiocephaly
Brief Title: Investigating the Effectiveness of Mobilization on Congenital Muscular Torticollis and Deformational Plagiocephaly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, Research Assistant, PhD, PT, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G014/14
Record Dates: First submitted 2015-03-15; First posted 2015-03-31 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Congenital Muscular Torticollis
Keywords: Congenital Muscular Torticollis; Manual Therapy; Infant
MeSH Terms: conditions — Congenital torticollis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soft tissue mobilization group (Experimental): soft tissue mobilization was applied three times in a week and home program exercises were recommended which consisted of positioning the neck and head, handling strategies, stretching exercises, strengthening exercises according to babies neurodevelopmental level and environmental adaptations
  Interventions: Other: soft tissue mobilization
- Home program controlled once six weeks (Experimental): Home program which consisted of positioning the neck and head, handling strategies, stretching exercises, strengthening exercises according to babies neurodevelopmental level and environmental adaptations were recommended
  Interventions: Other: home program controlled once six weeks

INTERVENTIONS:
Other: soft tissue mobilization — soft tissue mobilization technique has three phases. First phase 'the passive mobilization phase' is applied by gentle but tight gripping of the SKM muscle two or three fingers below the muscle origo and the muscle is mobilized rhythmically in the antero-posterior direction. Secondly, after gently continue to hold the muscle the baby was encouraged to do active repetitive cervical rotation to the affected side by means of catching the babies attention with colored and sonorous toys. Third phase was mobilization with stretching. Caregiver holds the baby on his/ her affected side while the therapist gently grips and withholds the muscle. Therapist mobilizes the muscle in the antero-posterior direction and stretch the muscle
  Arms: Soft tissue mobilization group
Other: home program controlled once six weeks — Home program which consisted of positioning the neck and head, handling strategies, stretching exercises, strengthening exercises according to babies neurodevelopmental level and environmental adaptations
  Arms: Home program controlled once six weeks

SUMMARY:
This study investigates the effect of soft tissue mobilization in babies with neck muscle problem. Babies received soft tissue mobilization or home exercises program

DETAILED DESCRIPTION:
Objectives: Investigating the effectiveness of soft tissue mobilization in babies with congenital muscular torticollis and deformational plagiocephaly.

Design: A Randomized controlled trial design Setting: University research department Participants:Babies with congenital muscular torticollis, aged between 0-6 months, who had a head tilt from 5 to 20 degrees and no other health problems were the participants of the study. The study included two groups; home program group was seen once every six weeks, the study group in addition to the home program also received soft tissue mobilization three times in a week. All groups received a baseline home program consisting of positioning, handling strategies plus stretching, stretching and strengthening exercises, environmental adaptations and classical massage. Babies were allocated to two groups by sealed envelope randomization. Babies were evaluated initially, at sixth weeks, at 12 weeks and follow-up at 18 weeks with muscle function scale, head tilt and ear shift assessments which included photographing method, neck normal range of motions (lateral flexion and rotation) and plagiocephaly severity scale

ELIGIBILITY:
Inclusion Criteria:

* Babies with congenital muscular torticollis and secondary deformational plagiocephaly
* Head tilt from 5 to 20 degrees
* Age between 0-6 months

Exclusion Criteria:

* Have another health problem such as neurological, vertebral anomalies, craniosynostosis

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Head tilt with photographic method | Change from Baseline in head tilt at 6th weeks of treatment, at the end of the treatment/12th weeks, at follow up/18th weeks
  Baby lies supine while taking photo of baby's habitual head position. The angle between the two lines, connecting eyes pupils and connecting acromions, is assessed.
plagiocephaly severity scale | Change from Baseline in at 6th weeks of treatment, at the end of the treatment/12th weeks, at follow up/18th weeks
  scale which has 5 subgroups as following frontal asymmetry, occipital flattening, head tilt, fascial asymmetry, ear asymmetry.

SECONDARY OUTCOMES:
Passive range of motion | Change from Baseline in at 6th weeks of treatment, at the end of the treatment/12th weeks, at follow up/18th weeks
  Baby lies in supine position and caregiver holds the baby's upper extremities by stabilizing shoulders to prevent compansatuar movements. For lateral flexion therapist bends the neck to opposite side from affected SCM. For neck rotation, therapist rotate the neck to affected SCM.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal KEKLİCEK, PhD,PT, Principal Investigator — Hacettepe University,Faculty of Health Sciences Department of Physiotherapy
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)